CLINICAL TRIAL: NCT04675866
Title: A Phase II Clinical Study of Camrelizumab Combined With Albumin-bound Paclitaxel and S-1 in the First-line Treatment of Advanced Gastric and Gastroesophageal Junction Adenocarcinoma
Brief Title: Camrelizumab Combined With Albumin-bound Paclitaxel and S-1 in the Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Houxinfang, Associate Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXGC-001
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-11

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — camrelizumab; Albumin-Bound Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab+albumin-bound paclitaxel+S-1 (Experimental): camrelizumab+albumin-bound paclitaxel+S-1
  Interventions: Other: Camrelizumab, Albumin-bound paclitaxel, S-1

INTERVENTIONS:
Other: Camrelizumab, Albumin-bound paclitaxel, S-1 — Camrelizumab: 200mg, iv, Q3W, d1; Albumin-bound paclitaxel: 125mg/m2, iv, d1, 8, Q3W; S-1: According to the patient's body surface area, the dosage is set to 40, 50, 60 mg/time, bid, po, taking 2 weeks, and stopping the drug for 1 week as a cycle.

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of Camrelizumab combined with paclitaxel (albumin binding type) and S-1 for first-line treatment of advanced gastric cancer, and to further explore the curative effect of PD - L1 expression in tumor tissue, EBV virus content, microsatellite instability (MSI), DNA mismatch repair (MMR), tumor mutation load (TMB), lymphocyte subgroup and cytokines.

DETAILED DESCRIPTION:
Gastric cancer is a common malignant tumor of digestive tract.The incidence of gastric cancer in China accounts for about half of the world's total, the incidence rate ranks second, and the mortality rate ranks second.Moreover, the proportion of early gastric cancer in China is very low, only about 20%. Most of them are in advanced stage at the time of discovery. The overall 5-year survival rate is less than 15%, which seriously threatens the health and life of Chinese people.For nearly 90% of HER2 negative patients with advanced gastric and gastroesophageal junction adenocarcinoma (g / GEJ), the current first-line treatment option is chemotherapy, and the efficacy of available drugs is very limited.The ORR of the first-line chemotherapy is about 40%, and the OS is about 10 months. New therapeutic drugs are urgently needed to improve the efficacy of advanced G/GEJ.The purpose of this study was to investigate the safety and efficacy of Camrelizumab combined with paclitaxel (albumin binding type) and S-1 for first-line treatment of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, no gender limit.
2. ECOG 0-1; estimated survival time ≥12 weeks.
3. Histopathologically confirmed unresectable locally advanced or metastatic HER-2 negative gastric adenocarcinoma.
4. At least one measurable lesion (RECIST1.1 standard).
5. Have not received systemic treatment for inoperable or metastatic gastric adenocarcinoma, past (new) adjuvant chemotherapy and adjuvant radiotherapy treatment ended to enrollment> 6 months.
6. For local lesions (non-target lesions) palliative treatment (mainly local radiotherapy) end time to random entry time> 2 weeks.
7. The main organs and bone marrow function are basically normal:

   1. Routine blood: neutrophils ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥80g/L;
   2. Liver function: TBiL≤1.5×ULN; ALT/AST≤2.5×ULN (for patients with liver metastases, ≤5ULN);
   3. Renal function: serum creatinine≤1.5×ULN and creatinine clearance rate>60mL/min;
   4. INR≤1.5×ULN and activated partial thromboplastin time ≤1.5×ULN.
8. Voluntary participation in the clinical study; fully understands and is informed of the study and has signed the Informed Consent Form (ICF); willing to comply with and able to complete all trial procedures.
9. Female subjects of childbearing age or male subjects whose sexual partners are females of childbearing age shall take effective contraceptive measures throughout the treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Patients with symptomatic central nervous system disease or meningeal metastasis; for patients with brain metastases who have received previous treatment, if the clinical condition is stable and imaging evidence does not show disease progression within 4 weeks before the first treatment, they can be considered for inclusion.
2. Patients who have previously been treated with albumin-bound paclitaxel or paclitaxel.
3. Received major surgery (craniotomy, thoracotomy or laparotomy), open biopsy or major traumatic injury within 28 days before enrollment, or expected major surgery during the study treatment period.
4. Suffered from other malignant tumors in the past 5 years (except for cured skin basal cell or squamous cell carcinoma, or carcinoma in situ such as cervix and breast).
5. The investigator believes that it will affect the subjects' ability to receive the treatment of the study protocol and are not controlled for serious medical diseases, such as combined serious medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, Active peptic ulcer, severe infection, etc.
6. Symptomatic congestive heart failure or cardiac color Doppler ultrasound examination shows LVEF (left ventricular ejection fraction <50%).
7. Any arterial thromboembolic events, including unstable angina pectoris and cerebrovascular accidents, occurred within 6 months before being selected for treatment.
8. A history of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism within 3 months before enrollment.
9. Participate in other clinical trials 28 days before enrollment, unless participating in observational (non-interventional) clinical research or in the follow-up phase of interventional research.
10. Patients with a history of interstitial lung disease, non-infectious pneumonia, or active tuberculosis.
11. Patients with congenital or acquired immune deficiency, active hepatitis B or C.
12. The patient is using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive purposes. Those who are still using it within 2 weeks before enrollment.
13. Patients with difficult-to-control effusion, accompanied by severe pleural effusion, abdominal effusion and other clinical symptoms.
14. Patients with grade ≥ 2 sensory or motor neuropathy; patients with peripheral neuropathy NCT-CTCAE ≥ 2.
15. People with a history of psychotropic drug abuse and unable to quit or patients with mental disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Defined as the proportion of patients with a documented complete response, and partial response (CR+PR).

SECONDARY OUTCOMES:
Disease control rate (DcR) | up to 2 years
  defined as the proportion of patients with complete response, partial response and disease stabilization (CR+PR+SD).
Overall survival (OS) | up to 2 years
  Defined as the date from random grouping to death from any cause.
Progression free survival (PFS) | up to 2 years
  Defined as the time betwween the onset of treatment and the observation of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Tumor Hospital, Luoyang, Henan, China

REFERENCES:
- [Derived] Wu C, Li S, Hou X. Camrelizumab plus albumin-bound paclitaxel and S-1 as first-line treatment for patients with human epidermal growth factor receptor 2-negative advanced gastric or gastroesophageal junction adenocarcinoma: a phase 2 trial. Front Immunol. 2026 Jan 2;16:1634502. doi: 10.3389/fimmu.2025.1634502. eCollection 2025. PMID 41550955